CLINICAL TRIAL: NCT04418687
Title: Does the Use of an Orthoglide Device Improve Patient Outcome, Following Total Knee Replacement
Brief Title: Use of the Orthoglide for Improved Patient Outcome Following Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambreen Chohan (Other)
Collaborators: Blackpool Victoria Hospital (Other)
Responsible Party: Sponsor-Investigator, Ambreen Chohan, Research Fellow, Sponsor-Investigator, University of Central Lancashire
Organization: University of Central Lancashire (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRAS 235931
Record Dates: First submitted 2020-03-15; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Knee Osteoarthritis; Physiotherapy; Intervention; Rehabilitation; Exercise
Keywords: Knee Osteoarthritis; Orthoglide; Knee exercises; KOOS; rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Group 1: Physiotherapy with Orthoglide
  Group 2: Physiotherapy only
Masking Description: Due to the nature of the study it was not possible to blind the participant to the treatment being received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy only (Active Comparator): Standard treatment post Total Knee Arthroplasty
  Interventions: Other: Physiotherapy only
- Physiotherapy + Orthoglide intervention (Experimental): Standard treatment post TKA, with additional Orthoglide device provided.
  Interventions: Device: Orthoglide

INTERVENTIONS:
Device: Orthoglide — Knee rehabilitation device.
  Arms: Physiotherapy + Orthoglide intervention
Other: Physiotherapy only — Physiotherapy only.
  Other Names: Physiotherapy
  Arms: Physiotherapy only

SUMMARY:
Total knee replacements are a common orthopaedic procedure undertaken at Blackpool Victoria Hospital. Following surgery patients are routinely seen by Physiotherapists who prescribe exercises to improve the range of movement and strength of the knee joint, thus aiding recovery. One of the key exercises prescribed involves the bending and straightening of the knee to improve range of movement. At this early stage of rehabilitation , due to weakness in the knee joint, reducing any resistance to this motion is beneficial. The Orthoglide device is designed to aid the patient in performing this movement by reducing the friction/resistance caused by the heel sliding against the bed. Currently this is achieved using a 'slider board' and placing a rolled up piece of fabric under the patients heel. The aim of this study is to investigate whether or not issuing an Orthoglide device to patients following total knee replacements improves functional outcomes reported by the patient at 6 weeks and 12 weeks post-surgery. Participants will be assigned to either receive an Orthoglide device and standard Physiotherapy or standard Physiotherapy alone. A series of patient reported outcome measures will be taken pre-surgery, 6 weeks post surgery and 12 weeks post surgery and the results compared.

DETAILED DESCRIPTION:
It is hypothesised that issuing an Orthoglide device following total knee replacement will improve patient reported outcomes. The null-hypothesis is that there is no correlation between the issuing of an Orthoglide device and improved patient reported outcome measures post total knee replacement.

The following outlines the various stages which the research participants will pass through during the study:

1. Initial contact - having been identified as requiring a total knee replacement the patient will attend Blackpool Victoria Hospital for a routine pre-operative assessment. During this contact the patient will be given an information pack relating to the project, this patient information sheet will include an invitation to participate, information regarding confidentiality, contact information as well as a consent form to be taken away and considered at home.
2. Homeward visit - The Homeward team routinely complete home visits with all patients who are awaiting a total knee replacement. During this visit the clinician will further discuss the study and, if the patient wishes to take part, the consent forms may be collected. The visiting clinician will store these sealed envelopes in-line with trust policy on data protection - in a lockable drawer/cabinet upon return to the hospital, this will only be accessible by the Homeward Team and research team.
3. Establishing baseline measurements - Consent forms will be reviewed by Robyn Jones and a copy placed in the patients records. Contact details will be recorded on secure access computer folder and participants contacted on preferred telephone number to establish baseline scores of outcome measures, gaining verbal consent prior to commencing. Consent forms will be stored in patients notes via coding with a further copy remaining in a secured storage location only accessible by the research team, for our records. Outcome measure scores will be inputted onto an anonymised and encrypted spreadsheet which will be stored on a password protected computer folder.
4. Randomisation - Due to the time period the trial will take place over the investigators will employ block randomisation to allow the participants to be grouped in a timely manner prior to their surgery. Once the participants identity has been anonymised and encrypted participants will be randomised in groups of 10, i.e. every 10 patients recruited will be randomised as one block. This process will repeat for every group of 10 recruited until capacity is reached for the intervention group and the control group. As a feasibility study it is estimated that 30 participants in each arm will be sufficient to give adequate power.
5. Identification of participants on weekly operation list - The Orthopaedic Physiotherapy team routinely access operation lists to identify the appropriate patients for Physiotherapy input. These operation lists will be cross referenced with our participant list to identify those taking part in the study and which group participants have been randomised into.
6. Patients will attend Blackpool Victoria Hospital for surgery. Routine post-operative Physiotherapy rehabilitation protocols will be followed with the only variation being the issue of an Orthoglide device to those in the study group and not to those in the control group - as identified in stage 5. Patients generally remain an in-patient for approximately 3 days post surgery.
7. 6 week follow up call - 6 weeks after the date of surgery (recorded in the secured spreadsheet from the weekly operation list)the research team will contact the patient to complete the outcome measures as used in stage 3, this data will be inputted onto the anonymised and encrypted spreadsheet stored on a password protected computer.
8. 12 week follow up call - 12 weeks after the date of surgery the research team will contact the patient to complete the outcome measures as used in stage 3 and 7, this data will be inputted onto the anonymised and encrypted spreadsheet stored on a password protected computer.
9. Data analysis and write up - Once all data is collected it will be analysed using the appropriate statistical analysis method and software. This study is designed to cause as little disruption to the routine patient journey as possible. Outside of routine contacts made by the direct care team, the only additional commitments participants must make is to be contacted by telephone by the research team 3 times (pre-operative baseline, 6 week follow-up and 12 week follow-up), each lasting approximately 20-15 minutes. It is estimated that from recruitment a participant will be involved with the study for a maximum of 24 weeks - preoperative clinics must be no more than 12 weeks prior to the surgery and the second follow-up phone call will be 12 weeks post operation. The overall timeframe for the project will be 24 months from April 2018 to April 2020, this includes ethics applications, data collection (to begin from November 2018), analysis and write up. Both arms of the trial will receive the same amount of Physiotherapy input (2 x daily visits) during their in-patient stay.

The only variable will be the issue of an Orthoglide device for the trial group to assist with completion of their knee exercises instead of a 'slider-board'. As a feasibility study no interim reports are planned however as soon as data has been analysed and reported upon it will be made available to the participants. participants will be randomised using block randomisation and data sets anonymised for analysis thus minimising researcher bias by all reasonable means for a study of this nature.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo a unilateral total knee replacement at Blackpool Victoria Hospital aged between 45 to 75 years,
* Independently mobile with or without a walking aid.

Exclusion Criteria:

* Other lower limb orthopaedic surgery within the last six-months,
* No anticipated further lower limb orthopaedic surgery within the next 12-months,
* No rheumatoid arthritis, neurological conditions affecting lower limb function.
* No Cognitive impairment,
* No co-morbidity which would act as a contraindication to engaging with prescribed exercise
* No existing participation in other clinical trials which may impact rehabilitation outcomes.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Knee Osteoarthritis Outcome Score (KOOS) | Change from Baseline to 6 and 12 weeks
  Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. A better score would be indicated by a higher number closer to 100.

SECONDARY OUTCOMES:
Change in Numerical Pain Rating Score (NPRS) | Change from Baseline to 6 and 12 weeks
  Scored from 0 to 10. Higher scores (closer to 10) indicate a higher level of pain and lower numbers indicate less pain. A minimal clinically important change in NPRS is a 2 point improvement.
Change in Exercise Adherence Rating Scale | Change from Baseline to 6 and 12 weeks
  EARS consists of 6 questions scored on a 5-point Likert scale, with positively worded questions reverse scored, giving a final rating from 0 (lowest adherence) to 24 (highest adherence). Better adherence is sought with any intervention

CONTACTS AND LOCATIONS:
Overall Officials: James Richards, PhD, Principal Investigator — University of Central Lancashire
Locations (1):
- Blackpool Victoria Hospital, Blackpool, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT04418687/ICF_000.pdf